CLINICAL TRIAL: NCT03105050
Title: Access to Bariatric Surgery In Europe
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: University College Dublin (Other); Sint Franciscus Gasthuis (Other); University Hospital, Ghent (Other); Lithuanian University of Health Sciences (Other); Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-0976
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: access; policy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Countries in Europe: All 51 countries will fill out their unique data on access to bariatric surgery in Europe
  Interventions: Other: Access to bariatric surgery

INTERVENTIONS:
Other: Access to bariatric surgery — All countries representatives will be interviewed on their Healthcare systems

SUMMARY:
In recent years more and more collaboration between hospitals performing bariatric surgery occur and more exchange of knowledge on pre and postoperative care is shared. Different countries have many different protocols to select and guide patients through bariatric surgery, and even within countries differences exist. These are most commonly based on expert opinions and cultural influences. Although many outcomes of the different approaches are known, the pathways the patient has to take and the accessibility to bariatric surgery are unclear for each country as well as how the care for these patients is financially arranged. As a progressive research collaboration, we would like to gain more insight into these different approaches. With this study we would like to gain more insight into the accessibility and restrictions to accessibility to both bariatric surgery and body contouring surgery after massive weight loss that exists in all 51 European countries, as well as why this disparity exists.

DETAILED DESCRIPTION:
Introduction

Bariatric surgery not only gives patients a new chance in life, but also facilitates improvements in social and mental status. Initially, guidance towards this life-changing surgery was often performed by the surgeons themselves. Before surgery, the patient had a short consultation and was given only limited information about the surgery and the expected results. The surgeon was often the only health care professional who made a judgment on whether a patient was suitable for bariatric surgery. On average, patients had annual or bi-annual postoperative follow-up. These visits focused in particular on weight loss and reduction in comorbidities. Today we know that this way of selecting and preparing patients for bariatric operations was inadequate. Many questions remained unanswered and patients did not know what to expect. In particular, many patients were unable to cope with the psychological adaptation required to undertake dietary and lifestyle changes to maximise weight loss. Because the number of follow-up visits were limited, many problems were not overcome.

There is a strong need for patients to have access to specialized professionals. In addition, it is very important to have patients screened by a multidisciplinary team before undergoing bariatric surgery. This team can quickly identify problems and can give advice on how to manage these. Although we all agree that morbid obese patients should have access to professional healthcare, we do not know the pathways the patient has to go to gain access. It seems logical that each country in Europe has his own pathways, but which one results in the best outcomes? As described above, there has been rapid growth in the number of patients undergoing bariatric surgery. Proper regulation of screening, follow-up and frequent counselling seems to strongly influence outcomes, like average weight loss. In the long term, a continuous supply of care is important to prevent weight gain. This has resulted in significant logistical issues for many hospitals, as care for each patient must be properly regulated and guaranteed. This care should be given for life, to identify and manage problems as quickly as possible.

In recent years more and more collaboration between hospitals occur and more exchange of knowledge on pre and postoperative care is shared. Different countries have many different protocols to select and guide patients through bariatric surgery, and even within countries differences exist. These are most commonly based on expert opinions and cultural influences. Although many outcomes of the different approaches are known, the pathways the patient has to take and the accessibility to bariatric surgery are unclear for each country as well as how the care for these patients is financially arranged. As a progressive research collaboration, we would like to gain more insight into these different approaches. With this study we would like to gain more insight into the accessibility and restrictions to access to both bariatric surgery and body contouring surgery after massive weight loss that exists in the different European countries, as well as why this disparity exists.

Research aim

To explore accessibility to bariatric surgery and quality of care in different European countries

Research objectives

1. To gain insight into the referral system for bariatric surgery in each European country for morbidly obese patients
2. To investigate the differences in inclusion criteria and registries for bariatric surgery per European country
3. To investigate the funding of bariatric and contouring surgery in each European country
4. To identify the differences in the multidisciplinary team providing care for bariatric patients
5. To identify the differences in the number of operations per surgeon and per hospital

In more detail:

1. Money:

   1. The amount of money which is used for reimbursement of bariatric surgery / Total amount of money in each healthcare system . This needs to be set in context with the population who does fulfil the criteria to undergo bariatric surgery according to (inter?)national guidelines.
   2. Methods to calculate reimbursement data: (Data from insurance companies: How much on average for a procedure? x Procedures (number and type) being performed a year (data from official register or society) per country
2. Guideline differences and Evidence)

   1. How does the country comply with the evidence and/or International Federation for Surgery on Obesity (IFSO) Consensus Statement?
   2. Are there specific national Guidelines?
   3. What are the criteria for reimbursement? Do they comply to national Guidelines?
3. Evaluation of the patient's journey:

   1. First contact to the bariatric surgeon... to bariatric surgery. (Differences in the system (self-referral, General Practitioner (GP) referral, etc.)
   2. Time interval from first contact to surgery
   3. Waiting time for elective surgery?
4. Quality:

   1. Patient collective (Are there differences? Baseline BMI / Co-morbidities?)
   2. Outcome (register: no register)
   3. How many patients undergo surgery in a centre
   4. How many patients undergo surgery in an University Hospital?
5. Plastic surgery

   1. How is referral arranged?
   2. Is it reimbursed and secondly how?

Methods

This study will be performed by the six researchers mentioned above. A questionnaire has been specifically designed for the purpose of this study (see appendix 1). Also, an inventory will be made as to who the national representatives for bariatric surgery are who can be interviewed.

The 51 countries have been divided between the six participants in this study and each participant will within six months gather the data required per country. Data will digitally be send to the research coordinator.

The IFSO secretary will be contacted to ask them to participate in this study and let us sent the questionnaire to all members. Secondly, the industry (Johnson and Johnson) will be asked to contact their connections on a nationwide scale to also sent the same questionnaire. If these are insufficient, we will try to contact insurance companies and/or patient groups to gain more data.

ELIGIBILITY:
Inclusion Criteria:

* Representative must be member of scientific community of his/her country for bariatric surgery
* All data of 2015 must be available for each country

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Representatives of bariatric communities per country in Europe
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Access to bariatric surgery per country (using a validated questionnaire) | 6 months
  Inventory accessibility
Quality of care per country (using a validated questionnaire) | 6 months
  Inventory quality of care

CONTACTS AND LOCATIONS:
Overall Officials: Yves van Nieuwenhove, MD, PhD, Study Chair — University of Gent; Almantas Maleckas, MD, PhD, Study Chair — Göteborg University
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will become available for other researchers in the form of articles, presentations and if requested